CLINICAL TRIAL: NCT07010315
Title: Development and Testing of a Patient-facing Educational Tool About Liver Cancer Prevention
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0299; NCI-2025-03535 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-05-09; First posted 2025-06-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Liver Cancer
Keywords: Liver cancer; Liver disease; Fibrosis; Cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Liver Diseases; Fibrosis | interventions — Neuropsychological Tests; User-Centered Design

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive Interviews (English and Spanish): Participants that agree to this part of the study will be asked to view patient education materials about liver cancer, complete a demographic survey, and do an interview one-on-one either online via Zoom, over the phone, or in person at HOPE Clinic.
  Interventions: Behavioral: Cognitive Testing
- Usability Testing (English and Spanish): Participants will be asked to complete a pre-survey, navigate a liver cancer education website, provide their feedback and impressions, and complete a post- survey.
  Interventions: Behavioral: Usability Testing

INTERVENTIONS:
Behavioral: Cognitive Testing — Given by Survey and one-on one interviews
  Groups: Cognitive Interviews (English and Spanish)
Behavioral: Usability Testing — Given by surveys and one-on-one interview.
  Groups: Usability Testing (English and Spanish)

SUMMARY:
To develop and test liver cancer prevention educational material.

DETAILED DESCRIPTION:
Primary Objectives:

* To ensure the text for the site is understood by participants, participant comprehension will be measured qualitatively through cognitive testing. Adjustments will be made to the content, messages, and layout iteratively until interviewer notes show no large discrepancies between participant understanding and the meaning of the text.
* To ensure the site is easy to use, usability will be measured qualitatively through usability testing. Adjustments will be made to the functionality of the patient-facing portions of the web-based tool iteratively until interviewer notes indicate that participants are able to input their risk factors and download the personal summary on their own.

Secondary Objectives:

* To describe whether the site is acceptable to users, acceptability will be measured (as part of usability testing) with the Ottawa Acceptability Measures.
* To describe participants' knowledge of liver cancer risk factors, knowledge will be measured (as part of usability testing) with Knowledge Questions developed for this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Participants at the HOPE Clinic
* Able to speak and read either English or Spanish
* For usability testing: Able to use and navigate websites on own smart phone or study computer

Exclusion Criteria:

* Has been diagnosed with liver cancer
* Cannot provide consent or otherwise participate in research activities (e.g. vision or hearing impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at HOPE Clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Testing | Up to 1.5 hours
  Participant comprehension will be measured qualitatively through cognitive testing. In cognitive testing interviews, participants are asked to "think aloud" as they review and react to new information. Participants will be presented with the storyboard (mock-up) versions of the content and asked to describe in their own words what the information means to them. Cognitive interviews may include questions about content such as length, clarity of the language, and helpfulness of the educational material. A trained research team member will ask probing questions throughout interviews as needed. Based on patient feedback, modifications will be made iteratively to the content to ensure the content is understood and interpreted as intended. There is no post-survey for cognitive testing.
Usability Testing | Up to 1.5 hours
  Usability will be measured qualitatively using a Usability Interview Guide. Usability will also be measured using the System Usability Scale. Acceptability will be measured with the Ottawa Acceptability Measures. Knowledge will be measured pre- and post- session using knowledge questions developed by the investigators and refined during cognitive testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hwang, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org